CLINICAL TRIAL: NCT01760629
Title: Hypothermia for Encephalopathy in Low Income Countries-Feasibility
Brief Title: Hypothermia for Encephalopathy in Low Income Countries-Feasibilty
Acronym: HELIX-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thayyil, Sudhin (Individual)
Collaborators: Government Medical College, Kozhikode (Other); Institute for Child Health, Madras Medical College, Egmore, Chennai (Unknown); Wayne State University (Other); Manipal Hospital, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3332/002
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Neonatal Encephalopathy
Keywords: Encephalopathy, Newborn, Low and Middle-income countries, Hypothermia
MeSH Terms: conditions — Brain Diseases; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cooling arm (Experimental): Whole body cooling to 33 to 34 C rectal temperature
  Interventions: Device: Tecotherm-HELIX

INTERVENTIONS:
Device: Tecotherm-HELIX — Whole body cooling using Tecotherm-HELIX
  Other Names: Therapeutic hypothermia; Whole body cooling

SUMMARY:
Whole body cooling improves survival with normal neurological outcome after neonatal encephalopathy in high-income countries. However, cooling equipments used in the high-income countries are expensive and unsuitable for wider use in low and middle-income countries (LMIC). We had previously conducted a randomised controlled trial of whole body cooling using phase changing material in south India. Although cooling was provided, there were wide temperature fluctuations.

Aim: To examine efficacy of the low technology cooling equipment (Tecotherm-HELIX) in administering effective and stable whole body cooling in encephalopathic infants.

Methods: After informed parental consent (and ethical approvals), we will administer 72 hours of whole body cooling (rectal temperature 33 to 34C) to a total 50 encephalopathic infants (aged <6 hours) admitted to the neonatal units at Calicut Medical College and Madras Medical College, over a six month period. To induce cooling, the infants will be kept on the cooling mattress. Temperature will be continuously measured for 80 hours using a rectal probe connected to a digital data logger.

The primary outcome will be the effective cooling time i.e. percentage of time (95% CI) for which the temperature remains between 33 to 340C during the intended cooling period.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 6 hours, Birth-weight >1.8, Gestation >36 weeks
2. Need for resuscitation at birth and 5 minute Apgar score <6 (in born babies) or Lack of cry by 5 minutes of age (for out-born babies)
3. Evidence of encephalopathy on clinical examination

Exclusion Criteria:

* Infants in moribound condition, where death is imminent
* Absent heart rate at 10 minute of age
* Major life threatening congenital malformation
* Lack of cooling equipment
* Lack of parental or physician consent

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of cooling | 72 hours
  To examine feasibility of whole body cooling within six hours of birth in infants with neonatal encephalopathy

SECONDARY OUTCOMES:
Short term morbidity | 2 weeks
  Short-term neonatal morbidity - Hypotension requiring inotropes, cardiac arrhythmias (other than bradycardia), coagulopathy/thrombocytopenia requiring blood products, respiratory failure requiring ventilatory support, seizures, and subcutaneous fat necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, PhD, Principal Investigator — Imperial College London; Seetha Shankaran, MD, Principal Investigator — Wayne State University, Michigan
Locations (3):
- India (3):
  - Manipal Hospital, Bangalore
  - Calicut Medical College, Calicut
  - Institute of Child Health, Madras Medical College, Chennai

REFERENCES:
- [Derived] Oliveira V, Kumutha JR, E N, Somanna J, Benkappa N, Bandya P, Chandrasekeran M, Swamy R, Mondkar J, Dewang K, Manerkar S, Sundaram M, Chinathambi K, Bharadwaj S, Bhat V, Madhava V, Nair M, Lally PJ, Montaldo P, Atreja G, Mendoza J, Bassett P, Ramji S, Shankaran S, Thayyil S. Hypothermia for encephalopathy in low-income and middle-income countries: feasibility of whole-body cooling using a low-cost servo-controlled device. BMJ Paediatr Open. 2018 Mar 23;2(1):e000245. doi: 10.1136/bmjpo-2017-000245. eCollection 2018. PMID 29637198